CLINICAL TRIAL: NCT06296329
Title: Rubber Hand Illusion in Anorexia Nervosa: the Role of Hand Dimensions and Physical Appearance
Brief Title: Rubber Hand Illusion in Anorexia Nervosa
Acronym: RHI_size_AN
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: University of Turin, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 21C309
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa
Keywords: bodily illusion; body representation
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Participants with Anorexia Nervosa
  Interventions: Other: Rubber Hand Illusion
- Controls: Not-hospitalized participants with a healthy weight
  Interventions: Other: Rubber Hand Illusion

INTERVENTIONS:
Other: Rubber Hand Illusion — The traditional behavioural illusion of the Rubber Hand will be applied

SUMMARY:
The present research project aims to verify a possible difference in the recalibration of the real hand position (i.e. proprioceptive drift) in relation to the dimensions of the plastic hand in the Rubber Hand Illusion, among a group of female participants with anorexia nervosa compared with a normal weight control group.

ELIGIBILITY:
Inclusion criteria:

* Right-handed
* diagnosis of Anorexia Nervosa according to the APA criteria

Exclusion criteria:

• concurrent neurological, neurodevelopmental (e.g., autism), motor, somatosensory and/or psychiatric disorders.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with anorexia nervosa will be recruited at the beginning of a rehabilitative treatment at the Istituto Auxologico Italiano, IRCCS, San Giuseppe Hospital (Italy). Controls will be recruited out of the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Proprioceptive drift in centimeters | baseline
  the recalibration of the real hand position towards the rubber hand

SECONDARY OUTCOMES:
Score at the Embodiment questionnaires | Baseline
  the score relative to the questionnaire measuring the individual experience towards the illusion. The higher is the score, the higher is the sense of illusion explicitely reported by participants.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Auxologico Italiano - Ospedale San Giuseppe, Piancavallo, VCO, Italy